CLINICAL TRIAL: NCT00470873
Title: A Non-Interventional, Post-Marketing Surveillance Phase IV Study to Obtain Data on Safety and Efficacy of Levitra® in Routine Treatment of Erectile Dysfunction in Depressive and Non-Depressive Men.
Brief Title: Vardenafil Treatment Of Erectile Dysfunction In Depressive And Non-Depressive Men
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 12842; LV0610PL; VALOR; NCT00459394 (obsolete NCT alias)
Record Dates: First submitted 2007-05-07; First posted 2007-05-08 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Levitra (Vardenafil, BAY38-9456)

INTERVENTIONS:
Drug: Levitra (Vardenafil, BAY38-9456) — Primary care erectile dysfunction patients for whom physician decided to start the treatment with vardenafil

SUMMARY:
The primary aim of this open, uncontrolled, prospective, non-interventional post-marketing surveillance study is to obtain data on safety and efficacy of Levitra in routine treatment of erectile dysfunction. The secondary aim of this study is to assess the influence of the treatment with Levitra on self-esteem (depressive symptomology) in men with ED.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Erectile dysfunction untreated or ineffectively treated with other than vardenafil PDE5 inhibitors

Exclusion Criteria:

* Treatment with nitrates
* Allergy to vardenafil or other tablets ingredients
* Treatment with CYP3A4 inhibitors (e.g. indinavir, ritonavir, ketoconazole, itraconazole, erythromycin)
* Cardiovascular status excluding any sexual activity

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care erectile dysfunction patients for whom physician decided to start the treatment with vardenafil
Sampling Method: Non-Probability Sample
Enrollment: 2471 (Actual)
Dates: Start 2007-01; Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Efficacy, safety, tolerance of the treatment with Vardenafil reported by the physician | At the patients control visit (approx. 3 months from the initial)

SECONDARY OUTCOMES:
Influence of vardenafil on depressive symptoms and self-esteem measured with CES-D and Rosenberg scale | At the patients control visit (approx. 3 months from the initial)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Poland